CLINICAL TRIAL: NCT01458392
Title: An Open-label Phase 2 Study of Dalantercept in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Study of Dalantercept in Patients With Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A041-03; dalantercept (Other: USAN)
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — ALK1-Fc fusion protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dalantercept (Experimental): dalantercept
  Interventions: Biological: Dalantercept

INTERVENTIONS:
Biological: Dalantercept — Subcutaneous dose of dalantercept once every 3 weeks.

SUMMARY:
Dalantercept, a soluble form of the activin receptor-like kinase-1 protein, is being studied in patients with squamous cell carcinoma of the head and neck (SCCHN). Dalantercept blocks the development of blood vessels that supply tumors.

DETAILED DESCRIPTION:
For cancer cells to grow, they need to have nutrients supplied to them through blood vessels. The study drug, dalantercept, is designed to work by blocking the growth of those blood vessels and preventing cancer cells from growing. The purpose of this study is to find out if dalantercept can cause SCCHN tumors to shrink or stop growing. This study will also evaluate the safety of dalantercept in patients with SCCHN.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically and/or cytologically confirmed, recurrent or metastatic SCCHN of mucosal origin (oral cavity, oropharynx, hypopharynx or larynx) not amenable to further local therapy (surgery, or radiation including re-irradiation); patients with unknown primary SCCHN presumed to be of head and neck mucosal origin are eligible if they meet all other entry criteria.
* Previously treated with at least one platinum-containing regimen or contraindicated for treatment with a platinum containing therapy. (Note: platinum therapy can occur upfront or after recurrence of disease. Failure of platinum therapy is not required.)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Key Exclusion Criteria:

* Nasopharyngeal carcinoma, paranasal sinus, salivary gland or primary skin SCCHN.
* Any other active malignancy for which chemotherapy or other anti-cancer therapy is indicated.
* Chemotherapy or other anti-cancer therapy or radiation therapy within 5 times the half-life of the drug or within 3 weeks prior to study day 1 if the half-life is not known.
* Treatment with another investigational drug or device, or approved therapy for investigational use, within 5 times the half-life of the drug or within 3 weeks prior to study day 1 if the half-life is not known.
* Major surgery within 4 weeks prior to study day 1 (patients must have recovered completely from any previous surgery prior to study day 1).
* Clinically significant cardiovascular risk.
* Clinically significant active pulmonary risk.
* Clinically significant active bleeding.
* Peripheral edema ≥ Grade 1 within 4 weeks prior to study day 1.
* Pregnant or lactating female patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Acceleron Investigative Site, Aurora, Colorado
  - Acceleron Investigative Site, Atlanta, Georgia
  - Acceleron Investigative Site, Boston, Massachusetts
  - Acceleron Investigative Site, Detroit, Michigan
  - Acceleron Investigative Site, New York, New York
  - Acceleron Investigative Site, Philadelphia, Pennsylvania
  - Acceleron Investigative Site, San Antonio, Texas
  - Acceleron Investigative Site, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Dalantercept 80 mg: Subcutaneous 80 mg dose of dalantercept once every 3 weeks.
- Dalantercept 0.6 mg/kg: Subcutaneous 0.6 mg/kg dose of dalantercept once every 3 weeks.
- Dalantercept 1.2 mg/kg: Subcutaneous 1.2 mg/kg dose of dalantercept once every 3 weeks.
Period: Overall Study
Arm/Group | Dalantercept 80 mg | Dalantercept 0.6 mg/kg | Dalantercept 1.2 mg/kg
Started | 2 | 13 | 31
Completed | 0 | 0 | 0
Not Completed | 2 | 13 | 31
Not completed — Death | 2 | 11 | 22
Not completed — At the discretion of the sponsor | 0 | 2 | 7
Not completed — Patient unwilling to comply with protoco | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalantercept 80 mg | Dalantercept 0.6 mg/kg | Dalantercept 1.2 mg/kg | Total
Number analyzed (Participants) | 2 | 13 | 31 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (13.4) | 59.6 (5.1) | 61.1 (9.5) | 60.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 5 | 7
  Male | 0 | 13 | 26 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 2 | 11 | 31 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 7 | 7
  White | 2 | 13 | 19 | 34
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 13 | 31 | 46

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the proportion of patients who met criteria for complete response or partial response. Patients were evaluable for ORR if they had at least one measurable lesion at baseline and at least one disease assessment after baseline. RECIST version 1.1 was used to evaluate efficacy. In addition, patients who developed clinical or radiological progression of disease prior to the scheduled tumor assessment were also considered evaluable for response. The response rate was estimated as the proportion of patients evaluable for response who meet the criteria for complete (CR) and partial response (PR). Per RECIST v1.1 for target lesions and assessed by MRI: complete response (CR), disappearance of all target lesions; partial response (PR), >=30% decrease in the sum of the longest diameter of target lesions; overall response (OR) = CR + PR.
Time Frame: Tumor assessments performed every 6 weeks, up to 30 days after the last dose of dalantercept and/or disease progression, up to approximately 2 years.
Population: The two patients at the 80 mg, fixed-dose level were excluded from the efficacy analysis as the protocol had been amended to incorporate weight-based dosing for the remainder of the study population. 40 received at least one dose of study drug in either the 0.6 mg/kg or 1.2 mg/kg dose groups and had at least one on-treatment tumor assessment.
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Dalantercept 0.6 mg/kg: Subcutaneous 0.6-mg/kg dose of dalantercept once every 3 weeks.
- Dalantercept 1.2 mg/kg: Subcutaneous 1.2-mg/kg dose of dalantercept once every 3 weeks.
Arm/Group | Dalantercept 0.6 mg/kg | Dalantercept 1.2 mg/kg
Number analyzed (Participants) | 13 | 27
participants | 0 [0 to 0] | 2 [0.9 to 24.3]

2. Secondary Outcome: Safety and Tolerability
Description: Number of participants with at least one adverse event as a measure of safety and tolerability.
Time Frame: Adverse events captured from first dose of dalantercept through 30 days after last dose of dalantercept.
Measure: Number; unit: participants
Arm/Group | Dalantercept 80 mg | Dalantercept 0.6 mg/kg | Dalantercept 1.2 mg/kg
Number analyzed (Participants) | 2 | 13 | 31
participants | 2 | 13 | 31

3. Secondary Outcome: Dalantercept Serum Concentration After Single and Multiple Doses
Description: Pharmacokinetic samples were collected pre- and post- dose on Days: 1, 8, 15, 22, 29, and 43. Reported below is AUC0-t (cycle 1).
Time Frame: Up to 43 days from initiation of treatment.
Population: The two patients at the 80 mg, fixed-dose level were excluded from the efficacy analysis as the protocol was amended to incorporate weight-based dosing for the remainder of the study population. 2 patients in the 0.6-mg/kg and 6 in the 1.2-mg/kg cohort had less than 2 measurable serum dalantercept concentrations and were excluded from PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*day/mL
Arm/Group | Dalantercept 0.6 mg/kg | Dalantercept 1.2 mg/kg
Number analyzed (Participants) | 12 | 26
ng*day/mL | 32992 (35.1) | 69572 (44.7)

4. Secondary Outcome: Dalantercept Serum Concentration After Single and Multiple Doses
Description: Pharmacokinetic samples were collected pre- and post- dose on Days: 1, 8, 15, 22, 29, and 43. Reported below is Cmax (cycle 1).
Time Frame: Up to 43 days from initiation of treatment.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dalantercept 0.6 mg/kg | Dalantercept 1.2 mg/kg
Number analyzed (Participants) | 12 | 26
ng/mL | 2446 (35.1) | 5336 (37.8)

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the date of the first dose to the first observation of disease progression (according to RECIST v.1.1) or death due to any cause. Progression is defined using RECIST v1.1 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: as for outcome 1
Population: The two patients at the 80 mg, fixed-dose level were excluded from the efficacy analysis as the protocol had been amended to incorporate weight-based dosing for the remainder of the study population.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Dalantercept 0.6 mg/kg | Dalantercept 1.2 mg/kg
Number analyzed (Participants) | 13 | 31
weeks | 5.8 [5.6 to 11.9] | 6.1 [5.7 to 11.7]

6. Secondary Outcome: Overall Survival (OS)
Description: OS is calculated as the number of months from date of the first dose to the date of death. The last patient treated will be followed for overall survival for 1 year following treatment initiation.
Time Frame: Survival captured until death or at a minimum 1 year from first dose of dalantercept.
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Dalantercept 0.6 mg/kg | Dalantercept 1.2 mg/kg
Number analyzed (Participants) | 13 | 31
weeks | 30.9 [13.6 to 45.6] | 41.3 [23.9 to 69.4]

7. Secondary Outcome: Disease Control Rate
Description: Disease control rate will be estimated as the proportion of patients evaluable for response who meet the criteria for complete response, partial response, or stable disease.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dalantercept 0.6 mg/kg | Dalantercept 1.2 mg/kg
Number analyzed (Participants) | 13 | 27
percentage of participants | 30.8 [9.1 to 61.4] | 44.4 [25.5 to 64.7]

ADVERSE EVENTS:
Arm/Group | Dalantercept 80 mg | Dalantercept 0.6 mg/kg | Dalantercept 1.2 mg/kg
Serious Adverse Events (participants affected / at risk) | 1/2 | 6/13 | 6/31
Other Adverse Events (participants affected / at risk) | 2/2 | 13/13 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalantercept 80 mg (N=2) | Dalantercept 0.6 mg/kg (N=13) | Dalantercept 1.2 mg/kg (N=31)
Tongue cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Disease progression (General disorders) | 0 | 1 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dalantercept 80 mg (N=2) | Dalantercept 0.6 mg/kg (N=13) | Dalantercept 1.2 mg/kg (N=31)
Fatigue (General disorders) | 1 | 8 | 12
Oedema peripheral (General disorders) | 0 | 2 | 11
Face oedema (General disorders) | 0 | 0 | 5
Oedema (General disorders) | 1 | 2 | 1
Pyrexia (General disorders) | 0 | 0 | 4
Malaise (General disorders) | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 2
Pain (General disorders) | 0 | 0 | 2
Catheter site pain (General disorders) | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dysphonia exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 4 | 11
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 4
Paresthesia (Nervous system disorders) | 0 | 1 | 3
Dizziness (Nervous system disorders) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 2 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 4
Vomiting (Gastrointestinal disorders) | 1 | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Tongue oedema (Gastrointestinal disorders) | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 16
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 9
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 3
Weight increased (Investigations) | 0 | 0 | 4
Weight decreased (Investigations) | 0 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2
Brain natriuretic peptide increased (Investigations) | 0 | 1 | 1
Lipase increase (Investigations) | 0 | 1 | 1
Blood urea increased (Investigations) | 0 | 1 | 0
Protein total decreased (Investigations) | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Feeding tube complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 3
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 1 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0
Macular degeneration (Eye disorders) | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 3
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No